CLINICAL TRIAL: NCT05307861
Title: Plastic vs Biodegradable Pancreatic Stent Comparison in the Prevention of Post-ERCP Pancreatitis: A Randomized Controlled Trial
Brief Title: Plastic vs Biodegradable Pancreatic Stent in Post-ERCP Pancreatitis Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IECED-14022022
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Biliary Tract Diseases
Keywords: Biliary tract diseases; pancreatic duct; stents
MeSH Terms: conditions — Biliary Tract Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pancreatic duct stenting with plastic stent (Active Comparator): Plastic pancreatic duct stent placement (5fr x 4 cm) for patients in need of pancreatic duct stenting during ERCP.
  Interventions: Device: Pancreatic duct stenting with plastic stent; Device: Pancreatic duct stenting with Biodegradable Stent
- Pancreatic duct stenting with Biodegradable Stent (Active Comparator): Biodegradable pancreatic duct stent placement (6fr x 4 cm or 6fr x 4 cm) for patients in need of pancreatic duct stenting during ERCP.
  Interventions: Device: Pancreatic duct stenting with plastic stent; Device: Pancreatic duct stenting with Biodegradable Stent

INTERVENTIONS:
Device: Pancreatic duct stenting with plastic stent — Plastic pancreatic duct stent placement (5fr x 4 cm) for patients in need of pancreatic duct stenting during ERCP.
Device: Pancreatic duct stenting with Biodegradable Stent — Biodegradable pancreatic duct stent placement (6fr x 4 cm or 6fr x 4 cm) for patients in need of pancreatic duct stenting during ERCP.

SUMMARY:
Multiple risk factors have been linked with post-endoscopic retrograde cholangiopancreatography pancreatitis (PEP); therefore, it is critical to follow strategies to reduce associated risk, morbidity, and mortality. However, there are also factors, such as pancreatic duct stenting, which have shown evidence of PEP prevention. The investigators pursue to compare plastic vs biodegradable pancreatic stents in the prevention of PEP.

DETAILED DESCRIPTION:
Endoscopic retrograde cholangiopancreatography (ERCP) is a high-skilled endoscopic procedure, which is currently mainly used as a therapeutic mean for various pancreaticobiliary disorders. Its most common serious adverse event is PEP. Multiple risk factors have been linked with PEP (patient/procedure/operator-related). Therefore, it is critical to follow strategies to reduce associated risk, morbidity, and mortality.

A recent metanalysis reported an overall incidence of PEP close to 10%, with an even higher incidence (14.7%) in high-risk patients. PEP's risk factors work synergically and have exhibited up to a 40% incidence rate in multifactorial patients. However, there are also factors, such as pancreatic duct stenting, which have shown evidence of PEP prevention.

The prophylactic use of pancreatic duct stents (especially 5 Fr stents) has exhibited a statistically significant PEP severity and incidence reduction; particularly for high-risk patients, for those who have undergone inadvertent repeated pancreatic duct cannulation or those in whom it is difficult to perform biliary cannulation. Controversially, failed pancreatic duct placement has shown a 34.7% PEP incidence rate and is considered an independent risk factor for PEP. In the case of stent migration, stent-induced perforation may arise regardless of the type of stent used (plastic or metallic), but if no signs of peritonitis are displayed, the endoscopic approach may suffice for stent removal and tracks closure. Rarely the surgical approach is guaranteed for migrated stents in the presence of peritonitis or retroperitoneal fluid collection.

The investigators pursue to compare plastic vs biodegradable pancreatic stents in the prevention of PEP.

ELIGIBILITY:
Inclusion Criteria:

* Patient is scheduled for ERCP
* Patient is 18 years old or older
* Biliary tract disease presence
* Non-manipulated pancreatic papilla
* Written informed consent provided

Exclusion Criteria:

* Patient not requiring pancreatic stenting during ERCP
* Failed pancreatic stent placement
* Patients at risk of fluid overload
* Patients with cholangitis, sepsis, acute/flared up chronic pancreatitis
* Recent previous biliary tract manipulation (i.e., pancreatoscopy, wirsungoscopy, etc.)
* Hemodynamic instability
* Uncontrolled coagulopathy, kidney/liver failure, or any comorbidity with a meaningful impact on cardiac risk assessment (NHYA III/IV)
* Pregnancy or nursing
* Refuse to participate in the study or to sign corresponding informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-01-30 (Estimated)

PRIMARY OUTCOMES:
PEP prevention at 72 hours | up to 72 hours after randomization
  Determine if plastic or biodegradable pancreatic stent placement renders PEP prevention. PEP is defined as proposed by Cotton et al in 1991(new hospitalization admission or 2/3-day hospital stay extension due to an abdominal pain suggestive of pancreatitis, plus a threefold increase of serum amylase/lipase above the normal limits 24 hours post-procedure).

SECONDARY OUTCOMES:
PEP prevention at 4 weeks | up to 4 weeks after randomization
  Determine if plastic or biodegradable pancreatic stent placement renders PEP prevention. PEP is defined as proposed by Cotton et al in 1991(new hospitalization admission or 2/3-day hospital stay extension due to an abdominal pain suggestive of pancreatitis, plus a threefold increase of serum amylase/lipase above the normal limits 24 hours post-procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Robles-Medranda, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Carlos Robles-Medranda, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ASGE Standards of Practice Committee; Chandrasekhara V, Khashab MA, Muthusamy VR, Acosta RD, Agrawal D, Bruining DH, Eloubeidi MA, Fanelli RD, Faulx AL, Gurudu SR, Kothari S, Lightdale JR, Qumseya BJ, Shaukat A, Wang A, Wani SB, Yang J, DeWitt JM. Adverse events associated with ERCP. Gastrointest Endosc. 2017 Jan;85(1):32-47. doi: 10.1016/j.gie.2016.06.051. Epub 2016 Aug 18. No abstract available. PMID 27546389
- [Result] Kochar B, Akshintala VS, Afghani E, Elmunzer BJ, Kim KJ, Lennon AM, Khashab MA, Kalloo AN, Singh VK. Incidence, severity, and mortality of post-ERCP pancreatitis: a systematic review by using randomized, controlled trials. Gastrointest Endosc. 2015 Jan;81(1):143-149.e9. doi: 10.1016/j.gie.2014.06.045. Epub 2014 Aug 1. PMID 25088919
- [Result] Freeman ML, Guda NM. Prevention of post-ERCP pancreatitis: a comprehensive review. Gastrointest Endosc. 2004 Jun;59(7):845-64. doi: 10.1016/s0016-5107(04)00353-0. No abstract available. PMID 15173799
- [Result] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Result] Moffatt DC, Yu BN, Yie W, Bernstein CN. Trends in utilization of diagnostic and therapeutic ERCP and cholecystectomy over the past 25 years: a population-based study. Gastrointest Endosc. 2014 Apr;79(4):615-22. doi: 10.1016/j.gie.2013.08.028. Epub 2013 Oct 8. PMID 24119510
- [Result] Mazaki T, Mado K, Masuda H, Shiono M. Prophylactic pancreatic stent placement and post-ERCP pancreatitis: an updated meta-analysis. J Gastroenterol. 2014 Feb;49(2):343-55. doi: 10.1007/s00535-013-0806-1. Epub 2013 Apr 24. PMID 23612857
- [Result] Buxbaum J, Yan A, Yeh K, Lane C, Nguyen N, Laine L. Aggressive hydration with lactated Ringer's solution reduces pancreatitis after endoscopic retrograde cholangiopancreatography. Clin Gastroenterol Hepatol. 2014 Feb;12(2):303-7.e1. doi: 10.1016/j.cgh.2013.07.026. Epub 2013 Aug 3. PMID 23920031
- [Result] Anderloni A, Fugazza A, Maroni L, Ormando V, Maselli R, Carrara S, Cappello A, Mangiavillano B, Omodei P, Preatoni P, Galtieri PA, Pellegatta G, Repici A. New biliary and pancreatic biodegradable stent placement: a single-center, prospective, pilot study (with video). Gastrointest Endosc. 2020 Aug;92(2):405-411. doi: 10.1016/j.gie.2020.02.049. Epub 2020 Mar 5. PMID 32145287
- [Result] Phillip V, Pukitis A, Epstein A, Hapfelmeier A, Haf D, Schwab M, Demir IE, Rosendahl J, Hoffmeister A, Schmid RM, Weber A, Algul H. Pancreatic stenting to prevent post-ERCP pancreatitis: a randomized multicenter trial. Endosc Int Open. 2019 Jul;7(7):E860-E868. doi: 10.1055/a-0886-6384. Epub 2019 Jul 3. PMID 31281872